CLINICAL TRIAL: NCT00375895
Title: Prospective, Open-label, Single Arm Pilot Study Evaluating the Effect on Virological Response of the Switch From Tacrolimus to Cyclosporin Associated With a Peginterferon Alfa-2a / Ribavirin Bitherapy, in Non-responder or With Recurrent VHC+ Disease Liver Transplanted Patients.
Brief Title: Switch From Tacrolimus to Cyclosporin in the Treatment of Recurrent Hepatitis C After Liver Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Rennes University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2006-002714-35; LOC/06-05 (Other: Rennes University Hospital); CIC0203/058
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Hepatitis C; Evidence of Liver Transplantation
Keywords: Cyclosporin; Peginterferon; Ribavirin; Chronic hepatitis C; Liver transplantation
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ciclosporin (Experimental)
  Interventions: Drug: ciclosporin

INTERVENTIONS:
Drug: ciclosporin — ciclosporin administered orally twice a day, at the initial dosing of 2.5 mg/kg/d, adjusted to obtain a C2 concentration of 600 ng/ml associated with the usual ribavirin and PEGinterferon bitherapy.
  Other Names: CsA; Cyclosporin

SUMMARY:
In France, 50% of hepatitis C virus carriers develop chronic clinical hepatitis, which may lead to cirrhosis and liver transplantation. Transplant infection by hepatitis C virus is constant after transplantation and recurrence causes chronic liver disease in 50 to 80% of cases. The aim of this study is to assess the efficacy of cyclosporin on C virological response. Patients included in the Transpeg 1 study and non-responder or with a recurrent disease will be switched from their tacrolimus therapy to cyclosporin, in association with a 1 year peginterferon alfa-2a / ribavirin bitherapy. Efficacy will be assessed by the percentage of patients with a negative qualitative PCR after 19 months of cyclosporin treatment.

DETAILED DESCRIPTION:
In France, 50% of hepatitis C virus carriers develop chronic clinical hepatitis, which may lead to cirrhosis and liver transplantation. Transplant infection by hepatitis C virus is constant after transplantation. A main factor determining the severity of recurrent hepatitis C after transplantation may be immunosuppression. Thus optimization of immunosuppressive regimens might be a key aspect to improve the prognosis of chronic hepatitis C in transplanted patients. The two most frequently used immunosuppressive drugs are cyclosporin and tacrolimus. However, it has been shown that virus replication could be inhibited by cyclosporin, through the blockade of cyclophilins, decreasing hepatitis C viral load and improving liver function. These effects were not found with tacrolimus.

The aim of our study is to assess the efficacy on C virological response of the switch from tacrolimus to cyclosporin associated with a peginterferon alfa-2a / ribavirin bitherapy, in non-responder or with a recurrent VHC+ disease liver transplanted patients.

Patients will receive a 19 month cyclosporin treatment, associated during 12 months with a peginterferon alfa-2a / ribavirin bitherapy. Efficacy will be assessed by the percentage of patients with a negative qualitative PCR after 19 months of cyclosporin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or over,
* Who had been included in the Transpeg 1 study,
* Non-responders after a three month peginterferon alfa-2a / ribavirin bitherapy or with a recurrent disease during the Transpeg 1 maintenance phase, whatever the randomization group (ribavirin or placebo),
* With a positive qualitative PCR at inclusion,
* With a METAVIR histologic score of 1 or more on the last biopsy (done within the 6 months preceding inclusion),
* Treated with tacrolimus for at least 6 months prior to inclusion,
* Having given a written informed consent.

Exclusion Criteria:

* Treatment with peginterferon or ribavirin within the 6 months preceding inclusion,
* Severe hepatocellular failure or decompensated cirrhosis,
* Acute graft rejection within the two months preceding inclusion, or signs of chronic rejection on the last biopsy, or retransplantation since inclusion in the Transpeg 1 study,
* Treatment with cyclosporin for more than 6 months during the 24 months preceding inclusion,
* Treatment with a mTOR inhibitor or with another investigational immunosuppressive drug,
* Positive serology for HIV or HBV,
* Cancer (or history of other malignancy during the last 5 years) except patients transplanted for hepatocellular carcinoma and basocellular or excised spinocellular carcinoma,
* Serious concomitant disease or acute or chronic disorder, other than the current transplant, treated with steroids,
* Serious cardiac pathology within the last 6 months,
* Women with ongoing pregnancy or breast-feeding,
* Serious chronic renal failure (creatinine clearance < 30 ml/mn),
* Haemoglobin < 10 g/dl, platelets < 50 000/mm3 or neutrophils < 1000 / mm3,
* Abnormal TSH values,
* Inability to cooperate or to communicate with the investigator,
* Contraindications to ribavirin, peginterferon alfa-2a or cyclosporin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Prolonged virological response | 19 months
  Percentage of patients with a negative qualitative PCR, 19 months after the initiation of cyclosporin treatment.

SECONDARY OUTCOMES:
Virological response 4, 7 and 13 months after the initiation of cyclosporin treatment | 4, 7 and 13 months
  Percentage of patient with negative or decreased quantitative PCR
Histological response: METAVIR score at 19 months | 19 months
Biological response: liver function at 4, 7, 13 and 19 months | 4, 7, 13 and 19 months
  Transaminases, gammaGT, alcalin phosphatase, total bilirubin.
Incidence of acute or chronic graft rejection at 19 months | 19 months
Incidence of death, graft loss and retransplantation at 13 and 19 months | 13 and 19 months
Renal function at 4, 7, 13 and 19 months | 4, 7, 13 and 19 months
  Creatinin clearance
Incidence of treatment discontinuation at 4, 7, 13 and 19 months | 4, 7, 13 and 19 months
Incidence of adverse events (cancers in particular). | 19 months

CONTACTS AND LOCATIONS:
Overall Officials: Yvon Calmus, MD, PhD, Principal Investigator — Hôpital Cochin, Paris; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (13):
- France (13):
  - Service d'Hépatologie - Hôpital Jean Minjoz, Besançon
  - Service d'Hépatogastroentérologie - Hôpital Beaujon, Clichy
  - Service d'Hépatologie et Gastroentérologie - CH Henri Mondor, Créteil
  - Service des Maladies de l'Appareil Digestif - CHRU Claude Huriez, Lille
  - Service de Chirurgie Générale - Hôpital Edouard Herriot, Lyon
  - Chirurgie Générale - Hôpital de la Conception, Marseille
  - Service d'Hépato-gastro-entérologie - Hôpital Saint Eloi, Montpellier
  - Chirurgie Viscérale et Digestive - Hôpital de l'Archet, Nice
  - Service de Chirurgie Générale - Hôpital Cochin, Paris
  - Service des Maladies du Foie - Hôpital Pontchaillou, Rennes
  - Service de Chirurgie Générale et Transplantation Multi-organe - Hôpital de la Hautepierre, Strasbourg
  - Service d'Hépato-gastro-entérologie - Hôpital de Rangueil, Toulouse
  - Centre Hépato-Biliaire - Hôpital Paul Brousse, Villejuif